CLINICAL TRIAL: NCT05156489
Title: An Open-Label, Interventional, Not Controlled Pilot Study to Assess Vestibular Mucosa Thickness by Ultrasound Evaluation and Vestibular Perception Thresholds Changes in Women Affected by Vestibulodynia (VBD) After One Cycle of Pixel CO2-Alma Fractionated Laser
Brief Title: Ultrasound Evaluation and Vestibular Perception Thresholds Changes in Women Affected by Vestibulodynia (VBD) After One Cycle of Pixel CO2-Alma Fractionated Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Filippo Murina (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor-Investigator, Dr. Filippo Murina, Head of the Pathology Service of the lower genital tract, ASST Fatebenefratelli Sacco
Organization: ASST Fatebenefratelli Sacco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDSV-2020-03.1
Record Dates: First submitted 2021-10-26; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Vestibulodynia (VBD) From at Least 6 Months
Keywords: Vestibulodynia (VBD); Fractionated Laser; Vaginal dryness.
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Intervention Model Description: Pilot open not comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fractionated Laser (Experimental)
  Interventions: Device: Fractionated Laser (Pixel CO2-Alma)

INTERVENTIONS:
Device: Fractionated Laser (Pixel CO2-Alma) — The Laser will be administered at baseline (visit 2, day 0), at visit 3 (day 28±4) and at visit 4 (day 56±4) into vestibule, following the IFU of the device.

SUMMARY:
Vestibulodynia (VBD), term revised by Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia in 2015, is a vulvar pain of at least 3 months' duration, without clear identifiable cause and localized at vestibuli.

Women affected by this disease report localized hypersensitivity and pain of the vulvar vestibule to the touch (eg, during sexual intercourse or tampon use). This pattern of responses is suggestive of sensory abnormalities in the form of evoked pain (eg, hyperalgesia or allodynia).

Research biopsy studies have demonstrated increased innervation of the vulvar vestibule and increased subepithelial heparinase activity and cytokines that have been associated with neuroinflammatory processes. In addition, the discomfort inherent in VBD is always associated with pelvic floor muscle overactivity, with the development of myofascial trigger points, resulting in localized or radiating pain and/or severe tenderness.

A rich nerve plexus was identified within the vaginal submucosa, which was only composed of sympathetic and parasympathetic axons, with contributions of smaller sensory fibers. The sensory nerve endings of the vulvar vestibule are dense and shallow, making this region more physiologically sensitive. Several works suggest that a thinner vestibular mucosa is more sensitive to nociception because nerve endings become more superficial, thus altering the transduction of mechanical pressure to facilitate nociception.

The CO2 fractionated laser, has been used to safely and effectively treat symptomatic vaginal atrophy. This tool has also been found to be useful in the treatment of vestibulodynia.

In this open pilot study, 30 female subjects aged more 18 years old at inclusion, having symptoms of VBD from at least 6 months, have given her informed consent and meet all the eligibility criteria, will be enrolled. The subjects will be treated with CO2 Fractionated Laser into vestibule, for 3 sessions at monthly intervals with a follow up of 4 months. Subjects will come to a total of 6 visits over a period of 3 months.

The primary objectives of the study are to evaluate the performance and safety of Pixel CO2-Alma Fractionated Laser in women affected by VBD by the assessment of vestibular mucosa thickness by ultrasound evaluation and vestibular perception thresholds changes at day 84 and 120 and by searching the adverse event during all the study. The secondary objectives are the assessment of VAS for burning/pain, and dyspareunia, evaluation of pain and hypersensitivity to the touch by Swab test, Female Sexual Function Index (FSFI) and by Vulval Pain Functional Questionnaire (VQ) at the visits.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by Vestibulodynia (VBD) from 6 months.
* Women older than 18 years and not yet in menopausa period (12 consecutive months without a menstrual period).
* Vulval pain from moderate to severe (in a Likert scale between 0 =absent and 10 =severe, scored at least 5 after sexual intercourse with penetration).
* Pain localized at vestibuli during sexual intercourse or in activities with pressure on vestibuli (ie bike, horsing).
* Willingness to provide informed consent
* Willing to have sexual intercourse in the study period

Exclusion Criteria:

* Hypersensitivity or intolerance to laser.
* Clinically significant findings on physical examination.
* Any chronic medical condition or psychologic disorder that per opinion of the Principal Investigator would make the patient ineligible for the study.
* Pelvic floor hypertonicity (from moderate to severe) evaluated at screening by the Investigator and scored on a Likert scale between 0 = hypertonicity absent and 3 =severe hypertonicity.
* Active vaginal or vulvar infections (e.g., herpes, candida, STIs)
* Uterine prolapse beyond the hymen.
* Subject has a history of scarring alteration (ie, keloid formation).
* Unknown past or active history of vaginal bleeding disorders.
* Any condition or behavior indicating to the Investigator that the subject is unlikely to be compliant with study procedures and visits.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women affected by Vestibulodynia (VBD)
Enrollment: 30 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Vestibular mucosa thickness measured in µm by B-scan ultrasonography (DermaScan C, Cortex Technology, Denmark) | 120 days
  The Investigator will use B-scan ultrasonography with a 20-MHz validated system. The changing was evaluated from baseline to day 84 (visit 5), and 120 (final visit).
Vestibular perception thresholds measured with values from 1 to 25 by Neurometer CPT (Neurotron, Inc, Baltimore, MD) | 120 days
  In Vestibular perception thresholds (VPT) a value ranging from 6 to 13 is classified as normal, while a value ranging from 1 to 5 show hyperesthesia. A value between 14 and 25 shows hypoesthesia.
  The changing was evaluated from baseline to day 84 (visit 5), and 120 (final visit).

SECONDARY OUTCOMES:
Dyspareunia by Visual Analogue Scale | 120 days
  The changing will be measured by Visual Analogue Scale (VAS) mean value from baseline to day 84 (visit 5), and 120 (final visit). The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms.
Burning/pain by Visual Analogue Scale | 120 days
  The changing will be measured by Visual Analogue Scale (VAS) mean value from baseline to day 84 (visit 5), and 120 (final visit). The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms.
Pain/hypersensitivity to the touch at Swab test measured by Visual Analogue Scale. | 120 days
  The changing from baseline to day 84 (visit 5), and 120 (final visit) will be reported in a Visual Analogue Scale (VAS). The minimum score is 0 and the maximum score is 10, where 0 represents no symptoms and 10 represents severe symptoms.
Sexual Function by Female Sexual Function Index | 120 days
  Sexual function will be evaluated at baseline and after 84 and 120 days by the Italian validated translation of the Female Sexual Function Index (FSFI), a self-report instrument consisting of 19 items that assess sexual function over the past 4 weeks in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. Mean value in each group separately and in the two groups in comparison will be analyzed.
Vulval pain by Vulval Pain Functional Questionnaire (VQ) | 120 days
  In the Vulval Pain Functional Questionnaire (VQ) a numerical value is assigned to each response. The higher the score the greater the functional limitation. A diminishing score represents improvement.
Vestibular trophism by the Vestibular Health Score | 120 days
  Vestibular Health Score (VHS) will be used by the Investigator evaluating 5 parameters (Petechiae, Pallor, Fragility, Dryness, Erythema) which lead to obtain a final score defining the degree of atrophy. Each item is scored on a Likert scale between 0 =absent and 3 =severe. Total scores range from 0 to 15.
Incidence of Treatment-Emergent Adverse Events/ Adverse Device Events/ Serious Adverse Events/ Serious Adverse Device Events [Safety and Tolerability] | up to 120 days
  The incidence will be calculated by searching for Adverse Event (AE), Adverse Device Event ADE, Serious Adverse Event (SAE), Serious Adverse Device Event (SADE) at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale dei Bambini "Vittore Buzzi", Milan, Italy

REFERENCES:
- [Background] Bornstein J, Goldstein AT, Stockdale CK, Bergeron S, Pukall C, Zolnoun D, Coady D; consensus vulvar pain terminology committee of the International Society for the Study of Vulvovaginal Disease (ISSVD); International Society for the Study of Women's Sexual Health (ISSWSH); International Pelvic Pain Society (IPPS). 2015 ISSVD, ISSWSH, and IPPS Consensus Terminology and Classification of Persistent Vulvar Pain and Vulvodynia. J Sex Med. 2016 Apr;13(4):607-12. doi: 10.1016/j.jsxm.2016.02.167. Epub 2016 Mar 25. PMID 27045260
- [Background] Goldstein AT, Pukall CF, Brown C, Bergeron S, Stein A, Kellogg-Spadt S. Vulvodynia: Assessment and Treatment. J Sex Med. 2016 Apr;13(4):572-90. doi: 10.1016/j.jsxm.2016.01.020. Epub 2016 Mar 25. PMID 27045258
- [Background] Wesselmann U, Bonham A, Foster D. Vulvodynia: Current state of the biological science. Pain. 2014 Sep;155(9):1696-1701. doi: 10.1016/j.pain.2014.05.010. Epub 2014 May 22. No abstract available. PMID 24858303
- [Background] Morin M, Binik YM, Bourbonnais D, Khalife S, Ouellet S, Bergeron S. Heightened Pelvic Floor Muscle Tone and Altered Contractility in Women With Provoked Vestibulodynia. J Sex Med. 2017 Apr;14(4):592-600. doi: 10.1016/j.jsxm.2017.02.012. PMID 28364981
- [Background] Farmer MA. What is special about the vulvar vestibule? Pain. 2015 Mar;156(3):359-360. doi: 10.1097/j.pain.0000000000000094. PMID 25687538
- [Background] Murina F, Barbieri S, Lubrano C, Cetin I. Vestibular Mucosa Thickness Measured by Ultrasound in Patients Affected by Vestibulodynia: A Case-Control Study. Sex Med. 2021 Apr;9(2):100320. doi: 10.1016/j.esxm.2020.100320. Epub 2021 Feb 13. PMID 33588370
- [Background] Salvatore S, Athanasiou S, Candiani M. The use of pulsed CO2 lasers for the treatment of vulvovaginal atrophy. Curr Opin Obstet Gynecol. 2015 Dec;27(6):504-8. doi: 10.1097/GCO.0000000000000230. PMID 26536212
- [Background] Murina F, Karram M, Salvatore S, Felice R. Fractional CO2 Laser Treatment of the Vestibule for Patients with Vestibulodynia and Genitourinary Syndrome of Menopause: A Pilot Study. J Sex Med. 2016 Dec;13(12):1915-1917. doi: 10.1016/j.jsxm.2016.10.006. Epub 2016 Nov 15. PMID 27864031